CLINICAL TRIAL: NCT03805347
Title: The Therapeutic Effect of Helminthostachys Zeylanica(L.)Hook on Functional Recovery After Surgical Operation in Patients With Ankle Fracture
Brief Title: The Therapeutic Effect of Dau-Di-Wu-Gong in Patient With Ankle Fracture
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 180917
Record Dates: First submitted 2019-01-04; First posted 2019-01-15 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Ankle Fractures
Keywords: Ankle fracture; Helminthostachys zeylanica(L.)Hook; Clinical trials; Functional recovery
MeSH Terms: conditions — Ankle Fractures | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Treatment group and Control group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication (Experimental): Extract of Helminthostachys zeylanica(L.)Hook in capsule, 1gm/time, 3 times daily
  Interventions: Drug: Helminthostachys zeylanica(L.)Hook
- Starch (Placebo Comparator): Starch in capsule，1gm/time, 3 times daily
  Interventions: Drug: Starch

INTERVENTIONS:
Drug: Helminthostachys zeylanica(L.)Hook — Extract of Helminthostachys zeylanica(L.)Hook, 1gm/time, 3 times daily
  Other Names: Dao-Di-Wu-Gong
  Arms: Medication
Drug: Starch — Starch in capsule, 1gm/time, 3 times daily
  Other Names: Placebo
  Arms: Starch

SUMMARY:
Ankle fracture is one of most common bone fracture in Taiwan, although ankle fracture can be treated by surgical operation, local edema, pain and wound poor healing always is noted, according to the investigator's knowledge, no good therapeutic methods to treat mention-above symptoms until now. Helminthostachys zeylanica(L.)Hook, also called Dau-Di-U-Gon has anti-inflammation, calm down heat and detoxication, and anti-edema. People in Taiwan often uses Helminthostachys zeylanica(L.)Hook to treat bone and tendon pain, and its Ugonin component of Helminthostachys zeylanica(L.)Hook also is proved that has analgesia and ant-inflammation. Therefore, the purpose of the present study was to design a randomized, double-blind, controlled study to evaluate functional recovery effect of Helminthostachys zeylanica(L.)Hook after surgical operation in patients with ankle fracture.

DETAILED DESCRIPTION:
the purpose of the present study was to design a randomized, double-blind, controlled study to evaluate functional recovery effect of Helminthostachys zeylanica(L.)Hook after surgical operation in patients with ankle fracture. The primary outcome measure was the scores change of American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot scale, and tape (figure-of-eight) methods. Secondary outcome measure was the level changes of bone metabolism in peripheral blood, four diagnostic method, and the changes of ankle X-ray findings.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 year-old male or female with acute ankle fractures with surgical indication (Joint line displacement >2mm ; fracture dislocation)

Exclusion Criteria:

* Previous skin disease, DM or peripheral vessel disease with local foot amputation.
* Previous ankle surgery, old ankle fracture, or open fracture.
* Liver or renal dysfunction, and cardiorespiratory failure.
* Surgical infection after surgery.
* Patient refuse or can't finish the treatment course
* Patient with cancer
* Pregnancy
* HIV positive.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Change of American Orthopedic Foot and Ankle(AOFAS) Score | 1st day of study, 10~14th days of study, 43th days of study
  Score to evaluate ankle and hindfoot function, from 0-100 points, healthy ankle 100 points
Change of Ankle volume | 1st day of study, 10~14th days of study, 43th days of study
  figure-of-8 method

SECONDARY OUTCOMES:
Level of bone turnover marker | 1st day of study, 43th days of study
  Alkaline Phosphatase(ALP)normal range between 37 and 116 U/L; type 1 procollagen amino-terminal-propeptide (P1NP), normal range between 20-42 ng/L
Fracture Healing | 1st day of study, 43th days of study
  ankle radiography, bone callus formation and continuity of callus

CONTACTS AND LOCATIONS:
Overall Officials: Ching Liang Hsieh, MD, PhD, Study Director — Graduate Institute of Integrated Medicine,China Medical University,Taiwan.; Lun Chien Lo, MD, PhD, Principal Investigator — School of Chinese Medicine,China Medical University,Taiwan.
Locations (1):
- ChangHua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YL, Shen CC, Shen YC, Chiou WF, Chen CC. Anti-inflammatory and Antiosteoporosis Flavonoids from the Rhizomes of Helminthostachys zeylanica. J Nat Prod. 2017 Feb 24;80(2):246-253. doi: 10.1021/acs.jnatprod.5b01164. Epub 2017 Feb 7. PMID 28169537
- See also: paper link — https://www.ncbi.nlm.nih.gov/pubmed/28169537